CLINICAL TRIAL: NCT02766257
Title: Anesthesia for Ambulatory Pediatric Surgery in Sub-Saharan Africa (SSA): a Pilot Study in Burkina Faso
Brief Title: Anesthesia for Ambulatory Pediatric Surgery in Sub-Saharan Africa (SSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Pédiatrique Charles de Gaulle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: A1
Record Dates: First submitted 2016-04-13; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Complications
MeSH Terms: interventions — Anesthesia

ARMS (1):
- children undergoing ambulatory surgery (Other)
  Interventions: Procedure: Anesthesia for ambulatory paediatric surgery

INTERVENTIONS:
Procedure: Anesthesia for ambulatory paediatric surgery

SUMMARY:
Long surgical wait-times and limited hospital capacity are common obstacles to surgical care in many countries in sub-Saharan Africa (SSA). Ambulatory surgery might offer a solution to these problems. The aim is to study the introduction of ambulatory surgery in a pediatric hospital in SSA.

This is a cross-sectional descriptive study which took place over 6 months. It includes all the patients assigned to ambulatory surgery in the Pediatric University Hospital in Ouagadougou, Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 status
* elective surgery with low potential for blood loss or severe pain, lasting less than 90 minutes
* whose parents could be contacted by telephone and who could return to the hospital in less than 1 hour
* Parents gave consent for the surgical procedure

Exclusion Criteria:

* non operative patients

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Failure of ambulatory surgery | 1day
  number of patients that have been hospitalized (for whom ambulatory have been conversed to hospitalization)

SECONDARY OUTCOMES:
Morbidity | 3 days
  Number of patients that presented complications of anesthesia or surgery such as nausea, vomiting, drowsiness and fever.
Complication after discharge from hospital | 3 days
  number of phone calls from parents of patients after ambulatory discharge

REFERENCES:
- [Derived] Kabre YB, Traore IS, Kabore FA, Ki B, Traore AI, Ouedraogo I, Bandre E, Wandaogo A, Ouedraogo N. Anesthesia for Ambulatory Pediatric Surgery in Sub-Saharan Africa: A Pilot Study in Burkina Faso. Anesth Analg. 2017 Feb;124(2):623-626. doi: 10.1213/ANE.0000000000001780. PMID 28067703